CLINICAL TRIAL: NCT02190994
Title: Effect of Perioperative Glucocorticoid Replacement on Prognosis of Surgical Patients With Sellar Lesions
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Shu Jiang, Professor Shu Jiang, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WestChina-2013137
Record Dates: First submitted 2014-07-05; First posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Pituitary Neoplasms; Craniopharyngiomas
Keywords: Hydrocortisone; Pituitary adenomas; Replacement therapy
MeSH Terms: conditions — Pituitary Neoplasms; Craniopharyngioma | interventions — Hydrocortisone; Prednisone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A. Normal function, non-GC replacement (No Intervention): No glucocorticoid replacement will be given perioperatively.
- B. Normal function, low-dose GC (Active Comparator): Hydrocortisone 100mg i.v. before anesthesia induction, and postoperative day 1. 80mg hydrocortisone at day 2; 60mg at day 3; 20mg at day 4; 5mg oral prednisone acetate tablet at day 4 and day 5; 2.5mg at day 6;
  Interventions: Drug: Hydrocortisone; Drug: Prednisone
- C. Impaired function, low-dose GC (Active Comparator): Hydrocortisone 100mg i.v. before anesthesia induction, and postoperative day 1. 80mg hydrocortisone at day 2; 60mg at day 3; 20mg at day 4; 5mg oral prednisone acetate tablet at day 4 and day 5; 2.5mg at day 6;
  Interventions: Drug: Hydrocortisone; Drug: Prednisone
- D. Impaired function, high-dose GC (Active Comparator): Hydrocortisone 100mg i.v. before anesthesia induction, and postoperative day 1 and day 2. 60mg hydrocortisone at day 3; 60mg at day 3; 20mg at day 4; 5mg oral prednisone acetate tablet per day, since postoperative day 3.
  Interventions: Drug: Hydrocortisone; Drug: Prednisone

INTERVENTIONS:
Drug: Hydrocortisone — used intravenously
  Arms: B. Normal function, low-dose GC; C. Impaired function, low-dose GC; D. Impaired function, high-dose GC
Drug: Prednisone — used as tablet form
  Arms: B. Normal function, low-dose GC; C. Impaired function, low-dose GC; D. Impaired function, high-dose GC

SUMMARY:
The purpose of this four-arm randomized controlled study is to determine whether eliminating glucocorticoids (GC) replacement in perioperative period in surgical patients with sellar lesion could result in similar or better outcomes comparing to traditional replacement therapy, regarding postoperative recovery of pituitary function and other postoperative complications (infection, pain, quality of life, recurrence). Surgical patients of our center with MRI-confirmed diagnosis of sellar lesion will be enrolled, insulin tolerance test (ITT) will be performed for assessment of the pituitary function at enrollment. Patients with normal pituitary function will be randomized into non-GC replacement group (group A) and low-dose GC replacement group (group B), while patients with impaired pituitary function will be randomized into low-dose GC replacement group (group C) and high-dose GC replacement group (group D). The primary outcome is the hypothalamic-pituitary-adrenal (HPA) -axis function of the patients, evaluated by plasma cortisol and adrenocorticotropic hormone (ACTH) levels. The secondary outcomes include the hypothalamic-pituitary-thyroid (HPT) axis function (TSH, thyroid-stimulating hormone, free T3, free T4), postoperative water-electrolyte balance, infection, recurrence and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Surgical patients with MRI-confirmed diagnosis of sellar lesions (non-functioning pituitary adenoma or craniopharyngioma)

Exclusion Criteria:

* Patients with pre-existing hyperthyroidism or Cushing's syndrome
* Patients with long-term glucocorticoids replacement history
* Patients with other co-morbidities that pose known influence upon the HPA-axis function (cardiovascular or cerebrovascular disease, metabolic disease or epilepsy)
* Patients with severe panhypopituitarism
* Patients with history of radiotherapy of the pituitary gland

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline plasma cortisol level | 1, 3, 5, 7, 30, 90, 180, 360 days post-op
  Plasma cortisol at 8:00, 16:00, 24:00 respectively
Change from baseline plasma ACTH level | 1, 3, 5, 7, 30, 90, 180, 360 days post-op
  ACTH at 8:00;
Change from baseline 24-hour urine free cortisol | 1, 3, 5, 7, 30, 90, 180, 360 days post-op
  24-hour urine free cortisol
Change from baseline insulin tolerance test result | 7, 30, 90 days post-op
  insulin tolerance test result

SECONDARY OUTCOMES:
Change from baseline plasma TSH level | 1, 3, 5, 7, 30, 90, 180, 360 days post-op
  plasma TSH level
Sodium, potassium concentration in the blood and urine | Daily post-op,for the duration of hospital stay, an expected average of 7 days
  Concentration of sodium, potassium in the blood and urine
Number of patients with postoperative infection | For the duration of hospital stay, an expected average of 7 days
  Routine blood test, body temperature fluctuation, cerebrospinal fluid test if necessary.
Change from baseline health-related quality of life | 7, 30, 90 days post-op
  The 15-Dimensions measure of health-related quality of life
Number of patients with recurred tumor | 3,6,12 months after surgery
  Enhanced MRI scan of the sellar region.
Change from baseline plasma free T3 level | 1, 3, 5, 7, 30, 90, 180, 360 days post-op
  plasma free T3 level
Change from baseline plasma free T4 level | 1, 3, 5, 7, 30, 90, 180, 360 days post-op
  plasma free T4 level
Urine output | Daily post-op,for the duration of hospital stay, an expected average of 7 days
  24-hour urine output

CONTACTS AND LOCATIONS:
Overall Officials: Shu Jiang, M.D., Principal Investigator — West China Hospital, Sichuan University, Chengdu, Sichuan, PR China
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China